CLINICAL TRIAL: NCT02493660
Title: A Prospective, Single Blinded, Multi-center, Randomized, Controlled, Pivotal Study to Assess the Safety and Effectiveness of the InSpace™ Device for Treatment of Full Thickness Massive Rotator Cuff Tears
Brief Title: A Pivotal Study to Assess the InSpace™ Device for Treatment of Full Thickness Massive Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoSpace Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLD-OR-010
Record Dates: First submitted 2015-07-01; First posted 2015-07-09 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Rotator Cuff Syndrome
Keywords: Massive Rotator Cuff Tear; Arthroscopy; Shoulder Joint; Rotator cuff partial repair

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- InSpace implantation (Experimental): Arthroscopic InSpace (Sub-acromial tissue spacer system) implantation
  Interventions: Device: InSpace sub-acromial tissue spacer system
- Tendon Repair (Active Comparator): Arthroscopic partial repair of rotator cuff
  Interventions: Procedure: Partial repair of rotator cuff

INTERVENTIONS:
Device: InSpace sub-acromial tissue spacer system — Arthroscopic implantation of InSpace sub-acromial tissue spacer system
  Arms: InSpace implantation
Procedure: Partial repair of rotator cuff — Arthroscopic partial repair of rotator cuff
  Arms: Tendon Repair

SUMMARY:
A pivotal study to assess the safety and effectiveness of the InSpace™ device implantation in comparison to surgical partial repair of full thickness Massive Rotator Cuff Tear (MRCT).

DETAILED DESCRIPTION:
This is a non-inferiority, prospective, single blinded, multi-center, randomized, controlled, pivotal study evaluating the safety and effectiveness of the InSpace™ device as a primary surgical treatment for full thickness MRCT in comparison to Partial Repair of a full thickness MRCT performed during an arthroscopic procedure.

ELIGIBILITY:
Main Inclusion Criteria:

* Positive diagnostic imaging by MRI of the index shoulder indicating a full thickness Massive Rotator Cuff Tear (MRCT), measuring ≥ 5 cm in diameter involving ≥ two tendons (confirmed Intra-operatively)
* Functional deltoid muscle and preserved passive range of motion on physical examination
* Documented VAS score of > 30 mm pain
* Failed non-operative treatment of at least 4 months
* Patient in general good health,independent, and can comply with all post-operative evaluations and visits.

Main Exclusion Criteria:

* Known allergy to the device material (copolymer of PLA and -ε-caprolactone)
* Evidence of the following conditions:

  1. significant gleno-humeral or acromiohumeral arthritis
  2. full thickness cartilage loss as seen on MRI
  3. gleno-humeral instability (excessive translation of the humeral head on the glenoid fossa)
  4. pre-existing deltoid defect or deltoid palsy
  5. major joint trauma, infection or necrosis
  6. partial thickness tears of the supraspinatous
  7. fully reparable rotator cuff tear [Tear of less than 5 cm in diameter (or < 4 cm2) with retractable tendon that can be fully repaired]
* The subject requires concomitant subscapularis repair and/or labral repair
* Previous surgery of the index shoulder in the past 1 year, excluding diagnostic arthroscopy
* The subject's condition is bilateral and rotator cuff repair is scheduled or to be scheduled over the course of this study for the contra lateral shoulder
* Major medical condition that could affect quality of life and influence the results of the study (e.g. HIV or other immunosuppressive conditions, active malignancy in the past 5 years, acute MI, CVA, etc.)
* Documented evidence of a history of drug/alcohol abuse within 12 months of enrollment
* The subject's condition represents a worker's compensation case
* The subject is currently involved in a health-related litigation procedure
* Females of child-bearing potential who are pregnant or breastfeeding or plan to become pregnant during the course of the study
* Concurrent participation in any other investigational clinical study one month prior to enrollment or during the entire study period
* The subject has implanted metallic devices (e.g., cardiac pacemakers, insulin pumps, nerve stimulators), medically implanted clips or other electronically, magnetically or mechanically activated implants that would contraindicate undergoing a MRI scan or has claustrophobia that would inhibit ability to undergo a MRI scan .
* The subject is physically or mentally compromised (e.g., currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, etc.), to the extent that the Investigator judges the subject to be unable or unlikely to remain compliant to follow-up
* The subject is receiving prescription narcotic pain medication for conditions unrelated to the index shoulder condition
* The subject currently has an acute infection in the area surrounding the surgical site.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Assaf Dekel, MD, Study Director — Ortho-Space
Locations (21):
- United States (18):
  - Southern California Orthopedic Institute, Van Nuys, California
  - University of Colorado, Denver, Colorado
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Midwest Orthopedics at RUSH, Chicago, Illinois
  - Rockford Orthopedic Associates, Rockford, Illinois
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - MedStar Union Memorial Orthopaedics, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - NYU, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Buffalo Buffalo, New York, New York
  - Upstate Orthopedics, Syracuse, New York
  - Cincinnati SportsMedicine and Orthopaedic Center - Mercy Health, Cincinnati, Ohio
  - The Ohio State University, Ohio City, Ohio
  - Rothman Institute, Philadelphia, Pennsylvania
  - University Orthopedic Center, State College, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Canada (3):
  - Fowler Kennedy Sport Medicine Clinic, London, Ontario
  - Roth McFarlane Hand and Upper Limb Center, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects assessed for eligibility n=229
Pre-assignment Details: Subjects excluded (n=45) for various reasons, not meeting criteria (n=11), declined to participate (n=12), and Other (n=22) such as, no medical clearance for surgery, intra-op screen failures, enrollment full.
Period: Overall Study
Arm/Group | InSpace Implantation | Tendon Repair
Started | 93 (ITT) | 91 (ITT)
Completed | 83 | 79 (Investigator requested subject be discontinued prior to any post-procedure efficacy assessments.)
Not Completed | 10 | 12
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Subject unable to return for follow-up visits | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Population: Number of subjects who were randomized and received an InSpace implant and the number of subjects who received a Partial Repair of their rotator cuff.
Groups:
- Total: Total of all reporting groups
Arm/Group | InSpace Implantation | Tendon Repair | Total
Number analyzed (Participants) | 93 | 91 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 44 | 82
  >=65 years | 55 | 47 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.8 (7.70) | 64.7 (7.88) | 65.8 (7.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 41 | 84
  Male | 50 | 50 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 91 | 89 | 180
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 83 | 80 | 163
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 12 | 27
  United States | 78 | 78 | 156

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in the Per Protocol Population With Surgical Treatment Success of the InSpace Device as a Primary Surgical Treatment for Full-thickness Massive Rotator Cuff Tears From Baseline to Month 12 With no SSSIs and no SADEs.
Description: The primary composite effectiveness endpoint was defined as achievement of improvement for the Western Ontario Rotator Cuff (WORC) score (≥275 points) and American Shoulder and Elbow Society (ASES) score (≥6.4 points) by week 6 and maintenance at month 12 without subsequent secondary surgical intervention (SSSI) or serious adverse device effects (SADEs).
  The improvement of points of the Western Ontario Rotator Cuff (WORC) of at least 275 (point scale of 0-2100:lower score is better) and American Shoulder and Elbow Society (ASES) at least 6.4 (point scale of 0-100:higher score is better) reflect the required number of points in improvement for treatment to be considered successful.
Time Frame: Baseline to month 12
Population: Percentage of participants in the Per Protocol Population (PP) with surgical treatment success of the InSpace device as a Primary surgical treatment for Full-thickness massive rotator cuff tears (MRCT).
Measure: Number; unit: percentage of participants
Arm/Group | InSpace Implantation | Tendon Repair
Number analyzed (Participants) | 88 | 88
percentage of participants | 51.1 | 39.8
Statistical Analysis 1: Comparison: InSpace Implantation vs Tendon Repair; Test type: Non-Inferiority — The non-inferiority margin was 10% for all composite endpoints. The primary analysis method was a multilinear regression model for month 12 success with age (<65 years, ≥65 years), gender, and treatment as the model covariates for the PP population for noninferiority testing; p = 0.0049, Regression, Logistic; Primary analysis method was for month 12 success with age (<65 years, ≥65 years), sex, and treatment as the model covariates

2. Secondary Outcome: Composite Endpoint of WORC Improvement ≥275 and ASES Improvement ≥6.4 at Week 6 Maintained at Month 24 no Subsequent Secondary Surgical Intervention (SSSI) and no Serious Adverse Device Effect (SADEs) (Pre-specified). Composite WORC ASES and Safety to M24
Description: Composite Endpoint Per Protocol Population (PP) of WORC Improvement ≥ 275 and ASES Improvement ≥ 6.4 from baseline at Week 6 Maintained at Month 24 with no Subsequent Secondary Surgical Intervention (SSSI) and no Serious Adverse Device Effect (SADEs) (pre-specified).
Time Frame: Baseline through to Month 24
Population: Per Protocol Population with no major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | InSpace Implantation | Tendon Repair
Number analyzed (Participants) | 82 | 79
percentage of participants | 46.3 [35.5 to 57.1] | 38.0 [27.0 to 49.0]

3. Secondary Outcome: Composite Endpoint Component Level Success for WORC at Month 12 Compared to Baseline in the Per Protocol Population (PP)
Description: The secondary effectiveness endpoint was defined as a composite component-level success at Month 12 for Western Ontario Rotator Cuff (WORC) total score improvement (≥275) (scale of 0-2100:lower score is better) in the two groups, InSpace and Partial Repair without subsequent secondary surgical intervention (SSSI) or serious adverse device effects (SADEs).
Time Frame: Baseline to month 12
Population: Per Protocol Population
Measure: Number; unit: percentage of participants
Arm/Group | InSpace Implantation | Tendon Repair
Number analyzed (Participants) | 88 | 88
percentage of participants | 89.8 | 87.5

4. Secondary Outcome: Composite Endpoint Component Level Success for ASES at Month 12 Compared to Baseline in the Per Protocol Population (PP)
Description: The secondary endpoint was defined as a composite component-level success for American Shoulder and Elbow Surgeons ( ASES) compared at baseline to Month 12 without subsequent secondary surgical intervention (SSSI) or serious adverse device effects (SADEs)..
  The total score improvement of (≥ 6.4 points) (scale of 0-100:higher score is better) from baseline in the two groups, InSpace and Partial Repair.
Time Frame: Baseline to month 12
Population: Per Protocol Population
Measure: Number; unit: percentage of participants
Arm/Group | InSpace Implantation | Tendon Repair
Number analyzed (Participants) | 88 | 88
percentage of participants | 96.3 | 90.9
Statistical Analysis 1: Comparison: InSpace Implantation vs Tendon Repair; Results from logistic regression model; Test type: Non-Inferiority — The non-inferiority margin was 10% for all composite endpoints; p < 0.05, Regression, Logistic

5. Secondary Outcome: Mean Change From Baseline to Month 24 in the Intent To Treat (ITT) Population With Available Data With Surgical Treatment Success of the InSpace Device as a Primary Surgical Treatment for Full-thickness Massive Rotator Cuff Tears Through to Month 24. WORC
Description: The secondary effectiveness endpoint was defined as mean change from baseline to Month 24 for Western Ontario Rotator Cuff (WORC) total score improvement (≥275) (scale of 0-2100:lower score is better) in the two groups, InSpace and Partial Repair.
Time Frame: Baseline through to month 24
Population: The Intent To Treat (ITT) population with available data.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | InSpace Implantation | Tendon Repair
Number analyzed (Participants) | 83 | 78
score on a scale | -1083.37 [-1199.94 to -966.81] | -1007.00 [-1108.34 to -905.67]

6. Secondary Outcome: Mean Change From Baseline to Month 24 in the Intent To Treat (ITT) Population With Available Data With Surgical Treatment Success of the InSpace Device as a Primary Surgical Treatment for Full-thickness Massive Rotator Cuff Tears Through to Month 24. ASES
Description: Mean change in American Shoulder and Elbow Surgeons (ASES) score from baseline to month 24.
  The improvement of points of the American Shoulder and Elbow Society (ASES) at least 6.4 (point scale of 0-100:higher score is better) reflect the required number of points in improvement for treatment to be considered successful.
Time Frame: Baseline through to month 24
Population: Intent To Treat (ITT) Population with available data
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | InSpace Implantation | Tendon Repair
Number analyzed (Participants) | 83 | 79
score on a scale | 46.22 [41.66 to 50.79] | 42.53 [37.96 to 47.10]

7. Secondary Outcome: Mean Change From Baseline to Month 24 for Constant-Murley (CS) in the Intent To Treat Population (ITT) With Available Data With Surgical Treatment Success of the InSpace Device as a Primary Surgical Treatment for Full-thickness Massive Rotator Cuff Tears
Description: The secondary effectiveness endpoint was defined as mean change from baseline to Month 24 for Constant-Murley (CS) Shoulder Outcome score (where the scale of 0-100:higher score is better) in the two groups, InSpace and Partial Repair.
Time Frame: Baseline to month 24
Population: Intent to Treat (ITT) Population with available data
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | InSpace Implantation | Tendon Repair
Number analyzed (Participants) | 83 | 79
score on a scale | 28.22 [23.92 to 32.51] | 21.81 [16.99 to 26.63]

8. Secondary Outcome: The Mean Change From Baseline to Month 24 for EQ-5D-5L for Intent To Treat (ITT) Population With Available Data With Surgical Treatment Success of the InSpace Device as a Primary Surgical Treatment for Full-thickness Massive Rotator Cuff Tears
Description: The secondary effectiveness endpoint was defined as change in baseline to Month 24 for Quality of Life (EQ-5D-5L) (scale of 0-100: lower score better) in the two groups, InSpace and Partial Repair.
Time Frame: Baseline through to month 24
Population: Intent to Treat (ITT) Population with available data
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | InSpace Implantation | Tendon Repair
Number analyzed (Participants) | 83 | 78
score on a scale | -4.65 [-5.36 to -3.94] | -4.00 [-4.61 to -3.39]

9. Secondary Outcome: Mean Change From Baseline to Month 24 for VAS in the Intent To Treat (ITT) Population With Available Data With Surgical Treatment Success of the InSpace Device as a Primary Surgical Treatment for Full-thickness Massive Rotator Cuff Tears
Description: The secondary effectiveness endpoint was defined as the mean change from baseline at Month 24 for Visual Analogue Scale (VAS) (scale of 0-100:lower score is better) in the two groups, InSpace and Partial Repair.
Time Frame: Baseline through to month 24
Population: Intent To Treat (ITT) Population with available data
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | InSpace Implantation | Tendon Repair
Number analyzed (Participants) | 83 | 78
score on a scale | -56.55 [-61.78 to -51.32] | -54.55 [-59.92 to -49.19]

10. Secondary Outcome: Mean Change From Baseline to Month 24 for ASES ROM in the Intent To Treat (ITT) Population With Available Data With Surgical Treatment Success of the InSpace Device as a Primary Surgical Treatment for Full-thickness Massive Rotator Cuff Tears
Description: The secondary effectiveness endpoint was defined as mean change from baseline at Month 24 for American Shoulder and Elbow Surgeons (ASES) range of motion (ROM)-physician reported portion. (scale of 0-180 Degrees: higher score is better) in the two groups, InSpace and Partial Repair.
Time Frame: Baseline through to month 24
Population: Intent to Treat (ITT) Population with available data
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | InSpace Implantation | Tendon Repair
Number analyzed (Participants) | 82 | 77
score on a scale | 36.89 [28.02 to 45.76] | 18.16 [9.33 to 26.98]

ADVERSE EVENTS:
Time Frame: Collected over 12 months and 24 months visit.
Description: The All-Cause Mortality, Serious Adverse Event, and Adverse events are listed for the safety population and some subjects reported more than one AE or SAE.
Arm/Group | InSpace Implantation | Tendon Repair
All-Cause Mortality (participants affected / at risk) | 0/93 | 1/91
Serious Adverse Events (participants affected / at risk) | 22/93 | 22/91
Other Adverse Events (participants affected / at risk) | 67/93 | 69/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InSpace Implantation (N=93) | Tendon Repair (N=91)
eg. Pain or inflammation (Musculoskeletal and connective tissue disorders) | 10 (11) | 11 (12) — All body areas reported
eg. dizziness, Aphasia, Cerebrovascular accident (Nervous system disorders) | 4 (6) | 2 (3)
eg.Prostate cancer, leukemia, Parathyroid tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 4 (4)
eg. Multi-vessel Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) — Same subject can have more than one event.
eg.Laryngeal granuloma, Chronic obstructive pulmonary disease, pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
eg. Gastrointestinal haemorrhage, short-bowel syndrome, small intestinal obstruction (Gastrointestinal disorders) | 2 (4) | 0 (0)
eg. Event leading to Death, non-cardiac chest pain, surgical failure (General disorders) | 0 (0) | 3 (3)
Angina Pectoris (Chest pain-Cardiac) (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Same subject can have more than one event.
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) — Same subject can have more than one event.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InSpace Implantation (N=93) | Tendon Repair (N=91)
Musculoskeletal pain, Arthralgia, back pain (anywhere in body) (Musculoskeletal and connective tissue disorders) | 51 (96) | 48 (71) — Note: One subject may have more than one event in all of these categories.
Fall and injury, meniscus injury, Tendon rupture (anywhere in body) (Injury, poisoning and procedural complications) | 13 (18) | 22 (23)
UTI, Bronchitis, pneumonia (Infections and infestations) | 16 (23) | 11 (13)
Headache, dizziness (Nervous system disorders) | 10 (14) | 10 (12)
Pain, Local swelling (General disorders) | 10 (12) | 5 (5)
Constipation (Gastrointestinal disorders) | 6 (10) | 6 (6)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) — Note: Some subjects may have more than one event.
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Pre-Ventricular Contractions (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of 45 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and can only extend the embargo with patent protection review.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT02493660/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT02493660/ICF_001.pdf